CLINICAL TRIAL: NCT06889181
Title: Evaluation of the Role of the Plasma-rich Growth Factor (PRGF) with Primary Cleft Palate Repair Versus Primary Cleft Palate Repair in Post-operative Wound Healing and Oronasal Fistula Occurrence, a Randomized Clinical Trial
Brief Title: Role of Plasma Rich Growth Factor in Repair Primary Cleft Palate
Acronym: PRGF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Samir Horia, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cleft palate - Omfs338
Record Dates: First submitted 2025-03-07; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cleft Palate; Plasma Rich in Growth Factors
Keywords: cleft palate; plasma rich growth factor; healing
MeSH Terms: conditions — Cleft Palate | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either control or study group in the ratio of 1:1 using random number table.
Who Masked: Participant
Masking Description: Single blinded study. Blinding to the patient will be ensured by masking the instruments during the follow up. The patient will be informed of the steps of the follow up (as mentioned in the consent form) without getting into details of the method of follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- plasma rich growth factor (PRGF) (intervention or study group) (Active Comparator): plasma rich growth factor (PRGF) intervention or study group Has Surgical procedures "von Langenbeck technique " to repair cleft palate and placing plasma rich growth factors between nasal and palatal tissue then primary closure intraoperatively, then patient will come for follow up visit after surgery, 1st day, 3rd, 5th day and come for follow up visits at 1 week, 1 month and 3 months postoperative
  Interventions: Other: Plasma Rich in Growth Factors (PRGF)
- placebo (control group) (Placebo Comparator): placebo (control group) Has Surgical procedures "von Langenbeck technique " to repair cleft palate primary closure, then patient will come for follow up visit after surgery, 1st day, 3rd, 5th day and come for follow up visits at 1 week, 1 month and 3 months postoperative
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Plasma Rich in Growth Factors (PRGF) — using prgf with closing primary cleft palate - isolated cleft palate Minutes before the surgery, 10-20 ml of venous blood from each patient. -The blood is centrifuged to obtain PRGF. -Fixed between nasal and palatal mucosa
  Arms: plasma rich growth factor (PRGF) (intervention or study group)
Other: Placebo — primary closing cleft palate-isolated cleft palate
  Arms: placebo (control group)

SUMMARY:
Does the plasma-rich growth factor (PRGF) with primary cleft palate repair accelerate wound healing and prevent post-operative oronasal fistula occurrence?

DETAILED DESCRIPTION:
The primary objective is to assess and evaluate the improvement of wound healing (edema at 5th day post operatively) as a primary outcome, and secondary objective is to assess and evaluate the wound closure and the decreasing of the occurrence of the oronasal fistula as a secondary outcome among children with cleft palate, using plasma rich growth factor between nasal mucosa and palatal mucosa

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients (American Society of Anesthesiologists -ASA I and II); not older than 6-18 months
* Patients with primary non-syndromic isolated cleft palate
* Apprehensive to be in the study.

Exclusion Criteria:

* Patients with recurrent palatal fistula
* Existence of syndromic cleft palate
* Blood diseases and platelet disorders (hematological disease)
* Systematic disease radiotherapy or chemotherapy for malignancy

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
wound healing assesment (edema at 5th day post operatively) | first day after surgery, 3rd day, and 5th day
  clinical records, percentage of persistence of edema number of participants with percentage of persisting of edema

SECONDARY OUTCOMES:
wound healing assesment | 2 years
  clinical records, counting days for healing as healing by days till closure
the occurrence of oronasal fistula | first day after surgery to end of treatment at 3 months
  clinical records, yes/no Postoperative complications; mainly oronasal fistula by; clinical observation: inspection, clinical signs: regurgitation of food or drink

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Manial, Cairo Governorate, Egypt